CLINICAL TRIAL: NCT07254468
Title: Effects of Cardiovascular Autonomic Neuropathy (CAN) on Acute Kidney Injury and Clinical Outcomes in Patients Undergoing Isolated Coronary Artery Bypass Surgery
Brief Title: Effect of Cardiovascular Autonomic Neuropathy on AKI and Outcomes in Isolated CABG Surgery
Acronym: CAN-AKI-CABG
Status: Active, not recruiting | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Emel Gunduz, Associate Professor of Anesthesiology, Akdeniz University, Antalya, Turkey, Akdeniz University
Other Study IDs: CAN_AKI_STUDY
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Acute Kidney Injury (AKI); Coronary Artery Bypass Graft (CABG); Cardiovascular Autonomic Neuropathy (CAN); Postoperative Outcomes
Keywords: Cardiovascular Autonomic Neuropathy (CAN); Acute Kidney Injury (AKI); Coronary Artery Bypass Graft (CABG)
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CABG Surgery Cohort: This cohort includes adult patients undergoing isolated coronary artery bypass graft (CABG) surgery with extracorporeal circulation (ECC). Each participant is evaluated preoperatively for cardiovascular autonomic neuropathy (CAN) using the Valsalva maneuver, sitting-to-standing test, and cold/heat test. Demographic, hemodynamic, and laboratory data, as well as regional cerebral oxygen saturation (rSO₂), are recorded. Postoperative outcomes include acute kidney injury (AKI) assessed by KDIGO criteria, complications, ICU and hospital stay, and mortality. No intervention is applied.

SUMMARY:
This study aims to investigate the effects of Cardiovascular Autonomic Neuropathy (CAN) on Acute Kidney Injury (AKI) and clinical outcomes in patients undergoing isolated Coronary Artery Bypass Graft (CABG) surgery requiring extracorporeal circulation(ECC).

Preoperative data including demographics, comorbidities, kidney function tests, hemodynamic parameters, and baseline regional cerebral oxygen saturation (rSO2) will be recorded. Intraoperative data will include hemodynamics, urine output, blood gases, cardiopulmonary bypass and aortic cross-clamp times, cardioplegia details, number of coronary anastomoses, and rSO2 changes at defined time points.

Postoperatively, kidney function, neurological status, mechanical ventilation duration, inotropic drug use, transfusion requirements, complications, ICU and hospital length of stay, and mortality will be evaluated. Acute Kidney Injury will be classified according to KDIGO criteria.

The primary objective is to analyze the effect of CAN on AKI. Secondary objectives include assessing the impact of CAN on other clinical outcomes and exploring the relationship between CAN and intraoperative cerebral oxygen changes.

This study has been approved by the Acıbadem University and Acıbadem Healthcare Institutions Medical Research Ethics Committee (ATADEK) and will be conducted following ethical principles and good clinical practice.

DETAILED DESCRIPTION:
This is a prospective, multicenter study investigating the effects of Cardiovascular Autonomic Neuropathy (CAN) on Acute Kidney Injury (AKI) and other clinical outcomes in adult patients undergoing isolated Coronary Artery Bypass Graft (CABG) surgery with planned extracorporeal circulation (ECC). The study aims to determine whether CAN is associated with AKI incidence and other postoperative outcomes.

Study Population:

Adults aged 18 years or older scheduled for elective isolated CABG surgery with planned ECC.

Inclusion Criteria:

Elective isolated CABG surgery Age ≥18 years

Exclusion Criteria:

Emergency or revision surgeries

Orthopedic conditions preventing standing tests

Chronic respiratory diseases affecting test reliability (COPD, asthma, chronic bronchitis)

Uncontrolled hypertension

Use of antiarrhythmic drugs affecting heart rate-based tests

Chronic kidney failure

Preoperative Assessment:

CAN diagnosis using Valsalva maneuver, sitting-to-standing test, and cold/heat test (positive if ≥2 tests are abnormal).

Collection of demographic data, comorbidities, laboratory tests (BUN, creatinine, GFR, ), hemodynamic parameters, and baseline regional cerebral oxygen saturation (rSO2).

Intraoperative Monitoring:

Hemodynamic parameters, urine output, blood gases, cardiopulmonary bypass and aortic cross-clamp times, and number of coronary anastomoses recorded.

Regional cerebral oxygen saturation (rSO2) continuously monitored during ECC, with values recorded for analysis but not used for clinical decisions.

Mean arterial pressure maintained at 60-100 mmHg; crystalloids infused at ≥100 ml/h; ephedrine administered if MAP <60 mmHg.

Postoperative Evaluation:

Kidney function monitored at 24h, 48h, and 7 days postoperatively using KDIGO criteria.

Evaluation of neurological outcomes, mechanical ventilation duration, inotropic support, transfusion requirements, postoperative complications (reoperation, mediastinitis, myocardial infarction), ICU and hospital length of stay, and mortality.

Study Objectives:

Primary: Assess the effect of CAN on AKI incidence.

Secondary: Evaluate CAN's impact on other clinical outcomes

Ethics and Compliance:

Approved by Acıbadem University and Acıbadem Healthcare Institutions Medical Research Ethics Committee (ATADEK), approval number 2020-21/13.

Conducted according to ethical principles and Good Clinical Practice (GCP) standards.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older

Scheduled for elective isolated Coronary Artery Bypass Graft (CABG) surgery with planned extracorporeal circulation (ECC)

Provide informed consent

Exclusion Criteria:Emergency or revision CABG surgeries

Chronic kidney failure or dialysis

Severe chronic respiratory disease (COPD, asthma, chronic bronchitis) affecting test reliability

Uncontrolled hypertension

Use of antiarrhythmic drugs affecting heart rate-based autonomic tests

Orthopedic or neurological conditions preventing standing tests

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients (≥18 years old) scheduled for elective isolated Coronary Artery Bypass Graft (CABG) surgery with planned extracorporeal circulation (ECC). Participants will be evaluated preoperatively for cardiovascular autonomic neuropathy (CAN) using standardized tests. Patients with chronic kidney failure, severe chronic respiratory disease, uncontrolled hypertension, or conditions preventing autonomic testing are excluded. Both male and female adults are eligible, and all participants must provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 884 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Kidney Injury (AKI) | Postoperative 7 days
  AKI will be assessed according to KDIGO criteria using serum creatinine, BUN, GFR values, and urine output within the first 7 days postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Faculty of Medicine, Department of Anesthesiology and Reanimation, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The data will be used solely for the purposes of this study."

REFERENCES:
- See also: Systematic review on the association between diabetic peripheral neuropathy and cardiac autonomic neuropathy. — https://doi.org/10.1016/j.jdiacomp.2024.108802

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT07254468/Prot_SAP_ICF_000.pdf